CLINICAL TRIAL: NCT02216214
Title: A Phase 4, Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multi-Center Study to Evaluate the Efficacy, Safety, and Tolerability of Mirabegron in Older Adult Subjects With Overactive Bladder (OAB)
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of Mirabegron in Older Adult Subjects With Overactive Bladder (OAB)
Acronym: PILLAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-MA-1005
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder (OAB)
Keywords: Urinary Incontinence; Mirabegron; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo to match mirabegron at an initial dose of 25 mg and may have been increased to 50 mg of matching placebo based on individual participant efficacy, tolerability and investigator discretion. Once a participant had increased dose, they remained on that dose for the remainder of the study unless there were safety reasons that required discontinuation of study drug.
  Interventions: Drug: Placebo
- Mirabegron (Experimental): Participants received mirabegron at an initial dose of 25 mg and may have been increased to 50 mg mirabegron after 4 weeks or 8 weeks based on individual participant efficacy, tolerability and investigator discretion. Once a participant had increased dose, they remained on that dose for the remainder of the study unless there were safety reasons that required discontinuation of study drug.
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — oral tablet
  Other Names: YM178; Myrbetriq
  Arms: Mirabegron
Drug: Placebo — oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the efficacy, safety and tolerability of mirabegron versus placebo in the treatment of older adult subjects with OAB.

ELIGIBILITY:
Inclusion Criteria assessed at Visit 1 (Screening):

* Subject is willing and able to complete the micturition diary and questionnaires correctly.
* Subject has symptoms of wet overactive bladder (OAB) (urinary frequency and urgency with incontinence) for greater than or equal to 3 months prior to Screening.
* Subject agrees not to participate in another interventional study from the time of screening until the final study visit.

Inclusion Criteria assessed after placebo run-in period at Visit 3 (Baseline):

* Subject continues to meet all inclusion criteria of Visit 1.
* Subjects must experience at least one incontinence episode in the placebo run-in period based on the 3-day micturition diary.
* Subject must experience at least 3 episodes of urgency (grade 3 or 4) based on the 3-day micturition diary.
* Subject must experience an average of greater than or equal to 8 micturitions/day based on the 3-day micturition diary.

Exclusion Criteria assessed at Visit 1 (Screening):

* Subject has ongoing symptoms suggestive of bladder outlet obstruction (BOO) or history of BOO that is currently not well controlled.
* Subject has Post-Void Residual Volume (PVR) greater than 150 mL.
* Subject has neurogenic bladder or neurological dysfunction or injury which could affect the lower urinary tract or nerve supply.
* Subject has significant stress incontinence or mixed stress/urgency incontinence where stress is the predominant factor as determined by the Investigator (for female subjects confirmed by a cough provocation test). Subjects with a history of stress incontinence that is currently treated (e.g. remote history of surgery for stress incontinence) may be included as long as they pass cough provocation test.
* Subject has an indwelling catheter or practices intermittent self-catheterization.
* Subject has evidence of Urinary Tract Infection (UTI). Urine culture and sensitivity will be performed for positive leukocytes, or nitrites, or turbidity, or at the investigator's discretion and will be confirmed with a culture greater than 100,000 cfu/mL. If a subject has a UTI at Screening (Visit 1), the subject can be rescreened after successful treatment of the UTI (confirmed by a laboratory result of negative urine culture).
* Subject has a chronic inflammatory condition such as interstitial cystitis, bladder stones, previous pelvic radiation therapy, or previous or current malignant disease of the pelvic organs (i.e., within the confines of the pelvis including the bladder and rectum in both sexes and the uterus, ovaries, and fallopian tubes in females; organs of the lower gastrointestinal tract are not necessarily considered pelvic organs as the distal ascending colon, the full transverse colon and proximal portion of the descending colon are in the abdomen).
* Subject resides in a nursing home.
* Subject is likely to enter a hospital or nursing home due to medical instability within the next 6 months in the opinion of the Investigator.
* Subject has received intravesical injection in the past 12 months with botulinum toxin, resiniferatoxin, or capsaicin.
* Subject has received electro-stimulation therapy for OAB (e.g. sacral nerve stimulation or Percutaneous Tibial Nerve Stimulation [PTNS]).
* Subject began or has changed a bladder training program or pelvic floor exercises less than 30 days prior to Screening.
* Subject has moderate or severe hepatic impairment defined as Child-Pugh Class B or C.
* Subject has severe renal impairment defined as estimated creatinine clearance less than 29 mL/min determined by Estimated Glomerular Filtration Rate (eGFR, Cockroft-Gault, or MDRD formulae). A subject with end stage renal disease or undergoing dialysis is also not a candidate for the study.
* Subject has severe uncontrolled hypertension, which is defined as a sitting systolic blood pressure greater than or equal to 180 mmHg and/or diastolic blood pressure greater than or equal to 110 mmHg.
* Subject has evidence of QT prolongation on electrocardiogram (ECG) defined as QTc greater than 450 msec for males, QTc greater than 470 msec for females or a known history of QT prolongation.
* Subject has a clinically significant ECG abnormality, as determined by the Investigator.
* Subject has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 2x upper limit of normal (ULN), or γ-GT greater than 3x ULN and considered clinically significant by the Investigator.
* Subject has a hypersensitivity to any components of mirabegron, other β-AR agonists, or any of the inactive ingredients.
* Subject has any clinically significant condition, which in the opinion of the Investigator makes the subject unsuitable for study participation.
* Subject has been treated with an experimental device within 28 days or received an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to Screening.
* Subject has a concurrent malignancy or history of any malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* Subject with current history of alcohol and/or drug abuse.
* Subject is using prohibited medications which cannot be stopped safely during the period.
* Subject has stopped, started or changed the dose of a restricted medication within the last 30 days prior to Screening.
* Subject is involved in the conduct of the study as an employee of the Astellas group, third party associated with the study, or the study site team.
* Subject has previously received mirabegron.

Exclusion Criteria assessed after placebo run-in period at Visit 3 (Baseline):

* Subject fulfills any exclusion criteria of Visit 1 (subject does not need to repeat screening assessments [PVR, cough provocation test, chemistry/hematology/urinalysis]).
* Subject was non-compliant during 2-week placebo run-in period, defined as taking less than 80% or greater than 120% of study medication.
* Subject has any systolic blood pressure measurement > 180 mmHg or diastolic blood pressure measurement > 110 in the 3-day diary or during the baseline visit.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 888 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc., Medical Affairs, Americas
Locations (120):
- United States (103):
  - Site US00066, Huntsville, Alabama
  - Site US00148, Mobile, Alabama
  - Site US00009, Anchorage, Alaska
  - Site US00020, Tucson, Arizona
  - Site US00019, Tucson, Arizona
  - Site US00063, Little Rock, Arkansas
  - Site US00081, Little Rock, Arkansas
  - Site US00176, Anaheim, California
  - Site US00048, Beverly Hills, California
  - Site US00142, Beverly Hills, California
  - Site US00150, Hawaiian Gardens, California
  - Site US00112, Los Angeles, California
  - Site US00034, Los Angeles, California
  - Site US00010, Murrieta, California
  - Site US00135, San Diego, California
  - Site US00139, San Diego, California
  - Site US00144, Santa Maria, California
  - Site US00083, Stanford, California
  - Site US00026, Colorado Springs, Colorado
  - Site US00039, Denver, Colorado
  - Site US00004, Denver, Colorado
  - Site US00040, New London, Connecticut
  - Site US00090, Washington D.C., District of Columbia
  - Site US00064, Brooksville, Florida
  - Site US00080, Coral Gables, Florida
  - Site US00002, DeBary, Florida
  - Site US00001, DeLand, Florida
  - Site US00017, DeLand, Florida
  - Site US00018, Edgewater, Florida
  - Site US00027, Fleming Island, Florida
  - Site US00151, Hialeah, Florida
  - Site US00179, Jupiter, Florida
  - Site US00057, Kissimmee, Florida
  - Site US00076, Lakeland, Florida
  - Site US00037, Miami, Florida
  - Site US00029, Miami, Florida
  - Site US00042, Miami, Florida
  - Site US00007, North Miami, Florida
  - Site US00021, Pompano Beach, Florida
  - Site US00035, Port Orange, Florida
  - Site US00075, St. Petersburg, Florida
  - Site US00099, Tampa, Florida
  - Site US00005, Savannah, Georgia
  - Site US00041, Boise, Idaho
  - Site US00060, Greenwood, Indiana
  - Site US00046, Jeffersonville, Indiana
  - Site US00134, West Des Moines, Iowa
  - Site US00104, Augusta, Kansas
  - Site US00105, Newton, Kansas
  - Site US00045, Overland Park, Kansas
  - Site US00172, Lake Charles, Louisiana
  - Site US00025, Annapolis, Maryland
  - Site US00091, Brockton, Massachusetts
  - Site US00006, New Bedford, Massachusetts
  - Site US00145, Watertown, Massachusetts
  - Site US00056, Grand Rapids, Michigan
  - Site US00003, Kalamazoo, Michigan
  - Site US00093, Saginaw, Michigan
  - Site US00024, Edina, Minnesota
  - Site US00137, Sartell, Minnesota
  - Site US00159, Billings, Montana
  - Site US00070, Norfolk, Nebraska
  - Site US00014, Las Vegas, Nevada
  - Site US00113, East Brunswick, New Jersey
  - Site US00111, New Brunswick, New Jersey
  - Site US00140, Albuquerque, New Mexico
  - Site US00016, Brooklyn, New York
  - Site US00043, Williamsville, New York
  - Site US00153, Charlotte, North Carolina
  - Site US00132, Concord, North Carolina
  - Site US00122, Greensboro, North Carolina
  - Site US00161, Raleigh, North Carolina
  - Site US00165, Wilmington, North Carolina
  - Site US00166, Winston-Salem, North Carolina
  - Site US00085, Fargo, North Dakota
  - Site US00067, Akron, Ohio
  - Site US00050, Cincinnati, Ohio
  - Site US00095, Cleveland, Ohio
  - Site US00084, Mentor, Ohio
  - Site US00015, Middleburg Heights, Ohio
  - Site US00102, Norman, Oklahoma
  - Site US00103, Portland, Oregon
  - Site US00180, Pittsburgh, Pennsylvania
  - Site US00082, Moncks Corner, South Carolina
  - Site US00162, Mt. Pleasant, South Carolina
  - Site US00032, Bristol, Tennessee
  - Site US00154, Chattanooga, Tennessee
  - Site US00053, Franklin, Tennessee
  - Site US00052, Nashville, Tennessee
  - Site US00175, Austin, Texas
  - Site US00131, Houston, Texas
  - Site US00174, Hurst, Texas
  - Site US00068, San Antonio, Texas
  - Site US00071, San Antonio, Texas
  - Site US00100, San Antonio, Texas
  - Site US00044, Salt Lake City, Utah
  - Site US00036, Salt Lake City, Utah
  - Site US00023, West Jordan, Utah
  - Site US00170, Newport News, Virginia
  - Site US00086, Norfolk, Virginia
  - Site US00167, Seattle, Washington
  - Site US00098, Tacoma, Washington
  - Site US00062, Madison, Wisconsin
- Canada (17):
  - Site CA00130, Edmonton, Alberta
  - Site CA00074, Vancouver, British Columbia
  - Site CA00155, Brampton, Ontario
  - Site CA00123, Corunna, Ontario
  - Site CA00169, Greater Sudbury, Ontario
  - Site CA00126, Hamilton, Ontario
  - Site CA00118, London, Ontario
  - Site CA00116, Sarnia, Ontario
  - Site CA00168, Toronto, Ontario
  - Site CA00164, Lévis, Quebec
  - Site CA00158, Montreal, Quebec
  - Site CA00073, Point Claire, Quebec
  - Site CA00106, Point Claire, Quebec
  - Site CA00156, Sherbrooke, Quebec
  - Site CA00061, Sherbrooke, Quebec
  - Site CA00129, Québec
  - Site CA00160, Québec

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Herschorn S, Staskin D, Schermer CR, Kristy RM, Wagg A. Safety and Tolerability Results from the PILLAR Study: A Phase IV, Double-Blind, Randomized, Placebo-Controlled Study of Mirabegron in Patients >/= 65 years with Overactive Bladder-Wet. Drugs Aging. 2020 Sep;37(9):665-676. doi: 10.1007/s40266-020-00783-w. PMID 32725584
- [Derived] Griebling TL, Campbell NL, Mangel J, Staskin D, Herschorn S, Elsouda D, Schermer CR. Effect of mirabegron on cognitive function in elderly patients with overactive bladder: MoCA results from a phase 4 randomized, placebo-controlled study (PILLAR). BMC Geriatr. 2020 Mar 18;20(1):109. doi: 10.1186/s12877-020-1474-7. PMID 32183741
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were ≥ 65 years who had symptoms of overactive bladder (OAB) were enrolled in 102 centers in 2 countries (US and Canada).
Pre-assignment Details: Eligible participants entered into a 2-week placebo run-in period. During this time, they were asked to complete a 3-day training micturition diary and in the 3 days prior to being randomized (and after, prior to each visit). Participants were randomized in a 1:1 ratio to either mirabegron or placebo, stratified by age (< 75 years, ≥ 75 years).
Groups:
- Placebo: Participants received placebo to match mirabegron at an initial dose of 25 mg and may have been increased to 50 mg of matching placebo after 4 weeks or 8 weeks based on individual participant efficacy, tolerability and investigator discretion. Once a participant had increased dose, they remained on that dose for the remainder of the study unless there were safety reasons that required discontinuation of study drug.
Period: Overall Study
Arm/Group | Placebo | Mirabegron
Started | 443 | 445
Treated | 442 | 445
Completed | 400 | 409
Not Completed | 43 | 36
Not completed — Randomized Never Received Study Drug | 1 | 0
Not completed — Adverse Event | 10 | 8
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 22 | 20
Not completed — Study Terminated By Sponsor | 0 | 1
Not completed — Miscellaneous | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): consisted of all randomized participants who received at least 1 dose of double-blind study drug. Participants from one site were excluded due to critical findings observed during a GCP audit of the site.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mirabegron | Total
Number analyzed (Participants) | 442 | 445 | 887
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (6) | 71.7 (5.5) | 71.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 324 | 317 | 641
  Male | 118 | 128 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 41 | 84
  Not Hispanic or Latino | 395 | 401 | 796
  Unknown or Not Reported | 4 | 3 | 7
Race [Count of Participants; unit: Participants]
  White | 357 | 348 | 705
  Black or African American | 25 | 33 | 58
  Asian | 54 | 59 | 113
  Other | 6 | 5 | 11
Age Categorical [Count of Participants; unit: Participants]
  < 75 years | 318 | 320 | 638
  ≥ 75 years | 124 | 125 | 249
Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: incontinence episodes/24 hours] — An incontinence episode was defined as the complaint of any involuntary leakage of urine. Population: Full analysis set-incontinence (FAS-I): included all participants who took at least 1 dose of double-blind study drug after randomization, reported at least 1 micturition and at least 1 micturition post-baseline and reported at least 1 incontinence episode in the baseline diary, and with available data and excluded participants from one site.
  incontinence episodes/24 hours
    number analyzed (Participants) | 430 | 437 | 867
    (all) | 3.44 (3.21) | 3.45 (3.11) | 3.44 (3.16)
Micturitions per 24 Hours [Mean (Standard Deviation); unit: micturitions/24 hours] — A micturition was defined as any voluntary act of passing urine (excluding incontinence only episodes). Population: The analysis population was the FAS-I, with available data.
  micturitions/24 hours
    number analyzed (Participants) | 430 | 437 | 867
    (all) | 10.5 (3.1) | 10.6 (2.4) | 10.6 (2.7)
Nocturia Episodes per 24 Hours [Mean (Standard Deviation); unit: nocturia episodes/24 hours] — A nocturia episode was defined as waking at night one or more time to void (i.e., any voiding associated with sleep disturbance between the date/time the participant goes to bed with the intention to sleep until the date/time the participant gets up in the morning with the intention to stay awake). A night time episode of incontinence only is not considered a nocturia episode. Population: The analysis population was the FAS-I, with available data.
  nocturia episodes/24 hours
    number analyzed (Participants) | 430 | 437 | 867
    (all) | 0.43 (0.71) | 0.45 (0.81) | 0.44 (0.77)
Urgency Episodes per 24 Hours (Grade 3-4) [Mean (Standard Deviation); unit: urgency episodes/24 hours] — An urgency episode was defined as the complaint of a sudden compelling desire to pass urine, which is difficult to defer, and is graded based on the Patient Perception of Intensity of Urgency Scale (PPIUS), where 3 = Severe urgency (I could not postpone voiding, but I had to rush to the toilet in order not to wet myself) and 4 =Urgency incontinence (I leaked before arriving to the toilet). Population: The analysis population was the FAS-I, with available data.
  urgency episodes/24 hours
    number analyzed (Participants) | 430 | 437 | 867
    (all) | 5.84 (3.87) | 5.88 (3.61) | 5.86 (3.74)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (EOT) in Mean Number of Micturitions Per 24 Hours
Description: A micturition was defined as any voluntary act of passing urine (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated as the average number of times a participant urinated per day during the 3-day micturition diary period.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: The analysis population was the FAS-I. Particpants with available data at baseline and EOT are included in the analysis. Last observation carried forward (LOCF) was used for EOT.
Measure: Least Squares Mean (Standard Error); unit: micturitions/24 hours
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 427 | 435
micturitions/24 hours | -1.7 (0.2) | -2.3 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Difference vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the ANCOVA model with treatment group, sex, age group (<75, >=75 years) and country as fixed factors and baseline value as a covariate; Test type: Superiority; p < 0.001, ANCOVA — P-value compares the Mirabegron group to the placebo group; Least Squares Mean (LSM) Mean Difference = -0.7, 95% CI 2-sided [-1.05 to -0.33], Standard Error of Mean 0.2

2. Primary Outcome: Change From Baseline to EOT in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated as the average number of times a participant recorded an incontinence episode per day during the 3-day micturition diary period.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: The analysis population was the FAS-I. Participants with available data at baseline and EOT are included in the analysis. LOCF was used for EOT.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes/24 hours
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 427 | 435
incontinence episodes/24 hours | -1.45 (0.13) | -2.00 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — P-value compares the Mirabegron group to the placebo group; LSM Difference = -0.55, 95% CI 2-sided [-0.82 to -0.27], Standard Error of Mean 0.14

3. Secondary Outcome: Change From Baseline to EOT in Mean Volume Voided Per Micturition
Description: The mean volume voided per micturition during 3 days of the 3-day micturition diary period.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 319 | 326
mL | 17.45 (4.17) | 30.54 (3.97)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Difference vs. Mirabegron: Differences of adjusted change from baseline values as well as the 95% CIs were generated from the stratified rank ANCOVA model with treatment group, sex, age group (<75, >=75 years) and country as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.002, stratified rank ANCOVA — P-value compares the Mirabegron group to the placebo group; LSM Difference = 13.68, 95% CI 2-sided [4.95 to 22.42], Standard Error of Mean 4.45

4. Secondary Outcome: Change From Baseline to EOT in Overactive Bladder Questionnaire (OAB-q): Symptom Bother Score
Description: The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQoL). The symptom bother portion consists of 8 questions, rated on a 6-point Likert scale (1 through 6). The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 (least severity) to 100 (worst severity). A negative change from baseline indicated an improvement.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 431 | 434
units on a scale | -18.69 (1.33) | -23.39 (1.29)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — P-value compares the Mirabegron group to the placebo group; LSM Difference = -5.15, 95% CI 2-sided [-7.84 to -2.46], Standard Error of Mean 1.37

5. Secondary Outcome: Change From Baseline to EOT in OAB-q: Health Related Quality of Life (HRQL) Total Score
Description: The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQoL). The HRQoL portion consists of 25 HRQoL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. The total score was calculated by adding the 4 HRQoL subscale scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 431 | 434
units on a scale | 14.80 (1.04) | 17.18 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.011, ANCOVA — P-value compares the Mirabegron group to the placebo group; LSM Difference = 2.72, 95% CI 2-sided [0.62 to 4.83], Standard Error of Mean 1.07

6. Secondary Outcome: Change From Baseline to EOT in Patient Perception of Bladder Condition (PPBC)
Description: The PPBC is a validated, global assessment tool using a 6-point Likert scale that asks participants to rate their subjective impression of their current bladder condition. Participants assessed their bladder condition using this scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems. A higher score indicated a worse perception of bladder condition.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 428 | 431
units on a scale | -0.7 (0.1) | -1.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — P-value compares the Mirabegron group to the placebo group; LSM Difference = -0.31, 95% CI 2-sided [-0.46 to -0.16], Standard Error of Mean 0.08

7. Secondary Outcome: Change From Baseline to EOT in Mean Number of Urgency Episodes (Grade 3 and/or 4) Per 24 Hours
Description: Urgency was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer. An urgency episode was defined as any micturition or incontinence episode with a severity of grade 3 or 4, assessed by participants based on the PPIUS, where 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could delay voiding a short while; 3 = Severe urgency, could not delay voiding; 4 = Urge incontinence, leaked before arriving to the toilet. The mean number of urgency episodes (grade 3 and/or 4) per 24 hours was calculated as the average number of times a participant recorded an urgency episode (grade 3 and/or 4) with or without incontinence per day during the 3-day micturition diary period.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: urgency episodes/24 hours
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 427 | 435
urgency episodes/24 hours | -2.81 (0.21) | -3.66 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Test type: Superiority; p < 0.001, ANCOVA — P-value compares the Mirabegron group to the placebo group

8. Secondary Outcome: Change From Baseline to EOT in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: An urgency incontinence episode was defined as the involuntary leakage of urine accompanied by or immediately preceded by urgency. The mean number of urgency episodes was calculated as the average number of times a participant recorded an urgency incontinence episode per day during the 3-day micturition diary period.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes/24 hours
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 427 | 435
urgency incontinence episodes/24 hours | -1.37 (0.12) | -1.93 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; The rate ratio for the number of urgency incontinence episodes reported during 3-day diary prior to each visit between mirabegron total group vs placebo group was calculated from a negative binomial regression model including treatment group, sex, age group (<75, >=75 years) and country as fixed factors and number of valid diary days as the offset variable; Test type: Superiority; p < 0.001, Negative Binomial Regression Model — P-value compares the Mirabegron group to the placebo group; Rate Ratio = 0.68

9. Secondary Outcome: Change From to EOT in Mean Number of Nocturia Episodes Per 24 Hours
Description: A nocturia episode was defined as waking at night one or more time to void (i.e., any voiding associated with sleep disturbance between the date/time the participant goes to bed with the intention to sleep until the date/time the participant gets up in the morning with the intention to stay awake). A night time episode of incontinence only is not considered a nocturia episode. The mean number of nocturia episodes per 24 hours was calculated as the average number of times a participant recorded a nocturia episode per day during the 3-day micturition diary period.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes/24 hours
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 427 | 435
nocturia episodes/24 hours | -0.21 (0.04) | -0.29 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; The rate ratio for the number of nocturia episodes reported during 3-day diary prior to each visit between mirabegron total group vs placebo group is calculated from a negative binomial regression model including treatment group, sex, age group (<75, >=75 years) and country as fixed factors and number of valid diary days as the offset variable; Test type: Superiority; p = 0.432, Negative Binomial Regression Model — P-value compares the Mirabegron group to the placebo group; Rate Ratio = 0.84

10. Secondary Outcome: Change From Baseline to EOT in Barthel Index of Daily Living Score
Description: The Barthel Index consists of 10 items that measure a person's daily functioning; specifically the activities of daily living and mobility. The total possible score ranges from 0 to 20, with lower scores indicating increased disability.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 415 | 420
units on a scale | 0.4 (0.1) | 0.5 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Test type: Superiority; p = 0.317, ANCOVA — P-value compares the Mirabegron group to the placebo group

11. Secondary Outcome: Change From Baseline to EOT in Vulnerable Elder Survey-13 (VES-13) Score
Description: The VES-13 is a simple function-based tool for screening community-dwelling populations to identify older persons at risk for health deterioration. The VES-13 considers age, self-related health, limitation in physical function, and functional disabilities. The total possible score ranges from 0 to 10, with higher scores indicating increased disability.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 177 | 176
units on a scale | -0.1 (0.1) | -0.3 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Test type: Superiority; p = 0.165, ANCOVA — P-value compares the Mirabegron group to the placebo group

12. Secondary Outcome: Change From Baseline to EOT in PPIUS
Description: The PPIUS is a 5-point categorical scale used by participants to rate the degree of associated urgency for each micturition and/or incontinence episode they experienced. categories include: 0 - No urgency, I felt no need to empty my bladder, but did so for other reasons; 1 - Mild urgency, I could postpone voiding as long as necessary, without fear of wetting myself; 2 - Moderate urgency, I could postpone voiding for a short while, without fear of wetting myself; 3 - Severe urgency, I could not postpone voiding, but had to rush to the toilet in order not to wet myself; 4 - Urge incontinence, I leaked before arriving at the toilet. Scores were recorded in the micturition diary.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 427 | 435
units on a scale | -0.37 (0.04) | -0.54 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Test type: Superiority; p < 0.001, ANCOVA — P-value compares the Mirabegron group to the placebo group

13. Secondary Outcome: Change From Baseline to EOT in OAB-q HRQL Subscale Scores
Description: The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQoL). The HRQoL portion consists of 25 HRQoL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. The Coping score has 8 items, the Concern score has 7 items, the Sleep and Social score has 5 items each. Each subscale score was calculated by adding each score's items and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicated an improvement.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 431 | 434
units on a scale
  Coping | 16.36 (1.23) | 18.95 (1.20)
  Concern | 16.89 (1.19) | 19.72 (1.16)
  Sleep | 13.46 (1.38) | 16.82 (1.35)
  Social | 11.15 (0.78) | 11.47 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Coping Subscale Score; Test type: Superiority; p = 0.019, ANCOVA — P-value compares the Mirabegron group to the placebo group
Statistical Analysis 2: Comparison: Placebo vs Mirabegron; Concern Subscale Score; Test type: Superiority; p = 0.010, ANCOVA — P-value compares the Mirabegron group to the placebo group
Statistical Analysis 3: Comparison: Placebo vs Mirabegron; Sleep Subscale Score; Test type: Superiority; p = 0.006, ANCOVA — P-value compares the Mirabegron group to the placebo group
Statistical Analysis 4: Comparison: Placebo vs Mirabegron; Social Subscale Score; Test type: Superiority; p = 0.614, ANCOVA — P-value compares the Mirabegron group to the placebo group

14. Secondary Outcome: Change From Baseline to EOT in Treatment Satisfaction Visual Analog Scale (TS-VAS)
Description: The TS-VAS is a visual analog scale that asks participants to rate their satisfaction with the treatment by placing a vertical mark on a line that runs from 0 (No, not at all) to 100 (Yes, completely).
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 427 | 429
units on a scale | 14.455 (2.058) | 20.110 (2.007)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Test type: Superiority; p = 0.002, ANCOVA — P-value compares the Mirabegron group to the placebo group

15. Secondary Outcome: Change From Baseline to EOT in University of Alabama, Birmingham - Life Space Assessment (UAB-LSA)
Description: The UAB-LSA measures mobility in terms of the spatial extent of a person's life. Life space is defined based upon the distance a person routinely travels to perform activities over this time frame. The UAB-LSA includes determining how far and how often the person leaves his or her place of residence and the degree of independence the person has. Each level of life space represents a distance further from the room where one sleeps: 0 - Mobility limited to the room where one sleeps; 1 - Mobility limited to within one's dwelling; 2 - Mobility limited to the space just proximal to one's personal living space (for instance, a porch, patio, or yard just outside the home or hallway outside of an apartment); 3 - Mobility limited to one's neighborhood; 4 - Mobility limited to one's town; 5 - Mobility outside one's town. The total scores ranges from 0-120, where a higher score indicates greater mobility.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 429 | 433
units on a scale | 1.33 (1.20) | 1.14 (1.17)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Test type: Superiority; p = 0.755, ANCOVA — P-value compares the Mirabegron group to the placebo group

16. Secondary Outcome: Change From Baseline in Number of Incontinence Episodes Reported During 3-Day Diary Prior to Each Visit
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The number of incontinence episodes were calculated as the total number of the incontinence episodes recorded during the 3-day micturition diary period.
Time Frame: Baseline and Weeks 4, 8 and EOT (up to 12 weeks)
Population: The analysis population was the FAS-I. Participants with available data at all time points are included in the analysis. LOCF was used for EOT.
Measure: Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 431 | 437
incontinence episodes
  Week 4: number analyzed (Participants) | 416 | 427
  Week 4 | -1.03 (0.12) | -1.44 (0.10)
  Week 8: number analyzed (Participants) | 406 | 404
  Week 8 | -1.36 (0.11) | -1.77 (0.11)
  EOT: number analyzed (Participants) | 427 | 435
  EOT | -1.40 (0.13) | -1.94 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Week 4: Rate ratio for the number of incontinence episodes reported during 3-day diary prior to each visit between mirabegron group vs placebo group is calculated from a negative binomial regression model including treatment group, sex, age group (<75, >=75 years) and country as factors and number of valid diary days as the offset variable; Test type: Superiority; p = 0.014, Negative Binomial Regression Model — P-value compares the Mirabegron group to the placebo group; Rate Ratio = 0.80, 95% CI 2-sided [0.67 to 0.96]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron; Week 8: Rate ratio for the number of incontinence episodes reported during 3-day diary prior to each visit between mirabegron group vs placebo group is calculated from a negative binomial regression model including treatment group, sex, age group (<75, >=75 years) and country as factors and number of valid diary days as the offset variable; Test type: Superiority; p = 0.043, Negative Binomial Regression Model — P-value compares the Mirabegron group to the placebo group; Rate Ratio = 0.81, 95% CI 2-sided [0.66 to 0.99]
Statistical Analysis 3: Comparison: Placebo vs Mirabegron; EOT: Rate ratio for the number of incontinence episodes reported during 3-day diary prior to each visit between mirabegron group vs placebo group is calculated from a negative binomial regression model including treatment group, sex, age group (<75, >=75 years) and country as factors and number of valid diary days as the offset variable; Test type: Superiority; p = 0.002, Negative Binomial Regression Model — P-value compares the Mirabegron group to the placebo group; Rate Ratio = 0.69, 95% CI 2-sided [0.54 to 0.87]

17. Secondary Outcome: Change From Baseline in Number of Pads During 3-Day Diary Prior to Each Visit
Description: The number of pads were calculated as the number of times a participant records a new pad used during the 3-day micturition diary period. No data were collected for the number of pads used due to a failure in the programming of the diary used for data collection.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: The analysis population was the FAS-I.
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Percentage of Participants Who Achieved Micturition Frequency Normalization
Description: Participants who achieved micturition frequency normalization were defined as participants who had at least 8 micturitions per 24 hours at baseline and less than 8 micturitions per 24 hours post-baseline.
Time Frame: End of treatment (up to 12 weeks)
Population: The analysis population was the FAS-I. Participants with available data at baseline and EOT are included in the analysis. Non-responder imputation (NRI) was used for EOT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 431 | 437
percentage of participants | 36.0 | 44.6
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Odds Ratio: Logistic regression was performed with treatment group, sex, age group (<75, >=75 years), and country as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.005, Regression, Logistic — P-value compares the Mirabegron group to the placebo group; Odds Ratio (OR) = 1.500

19. Secondary Outcome: Percentage of Participants With 50% Reduction in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. Participants with 50% reduction in mean number of incontinence episodes per 24 hours were defined as participants with at least 50% decrease from baseline in mean number of incontinence episodes per 24 hours during the treatment period at each visit.
Time Frame: End of treatment (up to 12 weeks)
Population: The analysis population was the FAS-I. Participants with available data at baseline and EOT are included in the analysis. NRI was used for EOT.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 428 | 435
percentage of participants | 60.0 | 72.4
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic — P-value compares the Mirabegron group to the placebo group; Odds Ratio (OR) = 1.775

20. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. Participants with zero incontinence episodes per 24 hours were defined as participants who had no incontinence episodes per 24 hours during the treatment period at each visit.
Time Frame: End of treatment (up to 12 weeks)
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 428 | 435
percentage of participants | 30.4 | 38.4
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.012, Regression, Logistic — P-value compares the Mirabegron group to the placebo group; Odds Ratio (OR) = 1.501

21. Secondary Outcome: Percentage of Participants With ≥ 10-Point Improvement From Baseline in OAB-q HRQL Subscales
Description: The OAB-q is a self-reported questionnaire with 33 questions relating to symptom bother and health-related quality of life (HRQoL). The HRQoL portion consists of 25 HRQoL items comprising 4 HRQoL subscales (Coping, Concern, Sleep, and Social Interaction), each item was scored 1-6. The Coping score has 8 items, the Concern score has 7 items, the Sleep and Social score has 5 items each. Each subscale score was calculated by adding each score's items and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. Participants with ≥ 10-point improvement from baseline in OAB-q HRQL subscales were defined as participants with at least 10-point improvement from baseline in OAB-q Subscales at each visit.
Time Frame: End of treatment (up to 12 weeks)
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 431 | 436
percentage of participants
  Coping | 58.7 | 66.1
  Concern | 56.6 | 62.2
  Sleep | 53.1 | 60.1
  Social | 34.1 | 36.9
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; HRQL Subscale - Coping. Odds Ratio: Logistic regression was performed with treatment group, sex, age group (<75, >=75 years), and country as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.034, Regression, Logistic — P-value compares the Mirabegron group to the placebo group; Odds Ratio (OR) = 1.390
Statistical Analysis 2: Comparison: Placebo vs Mirabegron; HRQL Subscale - Concern. Odds Ratio: Logistic regression was performed with treatment group, sex, age group (<75, >=75 years), and country as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.070, Regression, Logistic — P-value compares the Mirabegron group to the placebo group; Odds Ratio (OR) = 1.327
Statistical Analysis 3: Comparison: Placebo vs Mirabegron; HRQL Subscale - Sleep. Odds Ratio: Logistic regression was performed with treatment group, sex, age group (<75, >=75 years), and country as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.012, Regression, Logistic — P-value compares the Mirabegron group to the placebo group; Odds Ratio (OR) = 1.452
Statistical Analysis 4: Comparison: Placebo vs Mirabegron; HRQL Subscale - Social. Odds Ratio: Logistic regression was performed with treatment group, sex, age group (<75, >=75 years), and country as fixed factors and baseline value as a covariate; Test type: Superiority; p = 0.602, Regression, Logistic — P-value compares the Mirabegron group to the placebo group; Odds Ratio (OR) = 1.116

22. Secondary Outcome: Percentage of Participants With ≥ 1-Point Improvement From Baseline in PPBC
Description: The PPBC is a validated, global assessment tool using a 6-point Likert scale that asks participants to rate their subjective impression of their current bladder condition. Participants assessed their bladder condition using this scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems. A higher score indicated a worse perception of bladder condition. Participants with ≥ 1-point improvement from baseline in PPBC were defined as participants with at least 1-point improvement from baseline in PPBC at each visit.
Time Frame: End of treatment (up to 12 weeks)
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 428 | 433
percentage of participants | 54.4 | 64.7
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.001, Regression, Logistic — P-value compares the Mirabegron group to the placebo group; Odds Ratio (OR) = 1.634

23. Secondary Outcome: Percentage of Participants Major (≥ 2-Point) Improvement From Baseline in PPBC
Description: The PPBC is a validated, global assessment tool using a 6-point Likert scale that asks participants to rate their subjective impression of their current bladder condition. Participants assessed their bladder condition using this scale: 1. Does not cause me any problems at all; 2. Causes me some very minor problems; 3. Causes me some minor problems; 4. Causes me (some) moderate problems; 5. Causes me severe problems; 6. Causes me many severe problems. A higher score indicated a worse perception of bladder condition. Participants with ≥ 2-point improvement from baseline in PPBC were defined as participants with at least 1-point improvement from baseline in PPBC at each visit.
Time Frame: End of treatment (up to 12 weeks)
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 428 | 433
percentage of participants | 27.1 | 36.5
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.003, Regression, Logistic — P-value compares the Mirabegron group to the placebo group; Odds Ratio (OR) = 1.597

24. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety was assessed by AEs, which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. AEs were considered as serious if resulted in in death, was life-threatening resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly or birth defect, required inpatient hospitalization or led to prolongation of hospitalization and other medically important events.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 13 weeks)
Population: The analysis population was the SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 442 | 445
Participants
  AEs | 174 | 209
  Related AEs | 57 | 84
  AEs Leading to Deaths | 0 | 0
  SAEs | 12 | 15
  Drug-Related SAEs | 2 | 0
  AEs Leading to Study Drug Discont. | 14 | 14
  Drug-related AEs Leading to Study Drug Discont. | 7 | 10

25. Secondary Outcome: Change From Baseline to EOT in Montreal Cognitive Assessment (MoCA) Score
Description: The MoCA was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points, with lower scores indicating worse cognitive function.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: The analysis population was the SAF. Participants with available data at baseline and EOT are included in the analysis. LOCF was used for EOT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 411 | 425
units on a scale | -0.07 (0.14) | -0.16 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron; Test type: Superiority; p = 0.471, ANCOVA — P-value compares the Mirabegron group to the placebo group

26. Secondary Outcome: Change From Baseline in Post-void Residual Volume (PVR)
Description: PVR was assessed by ultrasonography or bladder scan.
Time Frame: Baseline and EOT (up to 12 weeks)
Population: The analysis population was the SAF. Participants with available data are included in the analysis. LOCF was used for EOT.
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Mirabegron
Number analyzed (Participants) | 380 | 377
mL | -3.1 (40.3) | 2.6 (56.2)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 13 weeks)
Arm/Group | Placebo | Mirabegron
All-Cause Mortality (participants affected / at risk) | 0/442 | 0/445
Serious Adverse Events (participants affected / at risk) | 12/442 | 15/445
Other Adverse Events (participants affected / at risk) | 12/442 | 23/445
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=442) | Mirabegron (N=445)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=442) | Mirabegron (N=445)
Headache (Nervous system disorders) | 12 (12) | 23 (23)

LIMITATIONS AND CAVEATS:
Participants from one site were excluded from the FAS-I and SAF due to critical findings observed during a GCP audit of the site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT02216214/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT02216214/SAP_001.pdf